CLINICAL TRIAL: NCT04427709
Title: Generate and Test the Reliability of a Pharmacodynamic Model of Oxytocin on Pupillary Hippus as a Measure of Central Nervous System Activity
Brief Title: Generate and Test the Reliability of a PD Model of OXT on Pupillary Hippus as a Measure of CNS Activity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00066475; 5P01NS119159-02 (NIH)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Osteoarthritis, Knee
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, crossover study. Each participant will receive Oxytocin 25 micrograms and placebo via intramuscular injection
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will be maintained by the research pharmacist and by an independent individual not affiliated with the data collection or outcome evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxytocin First, then Placebo (Other): Subjects in this arm will receive Intramuscular injection of Oxytocin (Pitocin®) first then placebo injection.
  Interventions: Drug: Oxytocin; Drug: Placebo
- Placebo, Then Oxytocin (Other): Subjects in this arm will receive Intramuscular placebo injection first then oxytocin injection
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intramuscular injection of Oxytocin (Pitocin®)
  Other Names: Pitocin
Drug: Placebo — Intramuscular placebo injection

SUMMARY:
The purpose of this research is to evaluate the effects of oxytocin (naturally occurring hormone) given by an intramuscular (IM; into the muscle) injection, has on your parasympathetic nervous system. The parasympathetic nervous system is the part of the involuntary nervous system that is sometimes called the "rest and digest" system; the parasympathetic system conserves energy as it slightly slows the heart rate, increases intestinal and gland activity, and relaxes sphincter muscles in the gastrointestinal tract.

DETAILED DESCRIPTION:
This is a single site study at Wake Forest School of Medicine. Healthy volunteers and patients with advanced knee arthritis being seen in the Orthopedic Clinic in consultation for potential total knee arthroplasty will be recruited after their doctor visit if the decision is made not to perform surgery at this time.

Study participants will come to the Pain Clinical Research Unit on 2 occasions. On these visits, they will receive an intramuscular (i.m.) injection of placebo or oxytocin, 25 micrograms (μg) (Pitocin®), obtained from the research pharmacy. The order in this cross-over study will be randomized and double blind, and the studies separated by at least 48 hours. Every 2.5 minutes beginning 20 minutes before injection and until 180 minutes after injection oscillation in pupil diameter at low frequency (hippus) will be obtained using an infrared pupilometer, in which they focus on a central point of gaze for 20 seconds. Hippus, a measure of parasympathetic output to the pupil and affected by central actions of oxytocin as described in preliminary data, will be calculated as the magnitude of power in the 0-0.25 Hertz (Hz) bin of the spectral analysis of pupil diameter, after removing blink and saccade artifacts. After 180 minutes the study participant will be discharged from the Pain Clinical Research Unit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3.
3. For healthy volunteers, normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication. For knee arthritis subjects, normal blood pressure or, for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.
5. Subjects with eye pathology, eye surgery, or taking topical eye medications, or any disease process that would cause motor tremors or excessive eye movements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fluctuation in Pupil Diameter (Hippus) -Pre drug administration | Baseline before study drug administration
  Magnitude of power at the dominant frequency in the Fourier transform of pupil diameter.
  One measure of coefficient of variation at each time period. It is calculated by the amount of variability in a window of time.
  Every 2.5 minutes beginning 20 minutes before the intramuscular injection of placebo or oxytocin, 25 micrograms.
Fluctuation in Pupil Diameter (Hippus) -Post drug administration | up to 180 minutes after study drug administration
  Magnitude of power at the dominant frequency in the Fourier transform of pupil diameter.
  One measure of coefficient of variation at each time period. It is calculated by the amount of variability in a window of time.
  Every 2.5 minutes for 180 after intramuscular injection of placebo or oxytocin, 25 micrograms.

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No